CLINICAL TRIAL: NCT05142644
Title: Intra Uterine Growth Retardation;Causes and Relationship
Brief Title: IUGR; Cause and Relationship
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Eva Wiberg-Itzel, Associate professor, Karolinska Institutet
Other Study IDs: Early or late IUGR
Record Dates: First submitted 2021-11-21; First posted 2021-12-02 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Intrauterine Growth Restriction
Keywords: IUGR; SGA
MeSH Terms: conditions — Fetal Growth Retardation | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early / growth restriction: Intrauterine growth restriction with onset before 32 weeks of gestation
  Interventions: Procedure: ultrasound
- Late growth restriction: Intrauterine growth restriction with onset after 32 weeks of gestation
  Interventions: Procedure: ultrasound

INTERVENTIONS:
Procedure: ultrasound — An extra ultrasound performed during pregnancy

SUMMARY:
Intrauterine growth restriction (IUGR) is a pregnancy complication in about 3-5% of all pregnancies in Sweden. IUGR fetuses are at high risk of morbidity and death. The method used in Sweden to detect IUGR is repeated measurements of pregnant women's symphysis-fundus measure (SF measure).

Weight estimation with ultrasound is performed only on indication; stagnant or deplaning SF dimensions or in the event of complications. Only high-risk pregnancies have repeated growth checks during pregnancy from the beginning.

There are potential benefits to detecting IUGR fetuses during pregnancy. Still, the effect is questioned. A meta-analysis of randomized studies could not benefit from a routine ultrasound in the third trimester.

The scientific purpose of this work is to evaluate the benefits of early detection and care of SGA (small for gestational age)/IUGR (growth-inhibited) fetuses and, if possible, to increase knowledge about this patient group. The hope is that this will lead to a better opportunity to personalize both preventive care and treatment of these women and children.

DETAILED DESCRIPTION:
Design: Register-based cohort study. Population: All pregnancies in Stockholm from 2014 to 2017 A Composite outcome for the study is constructed and consists of at least one of the following outcomes

1. HIE (hypoxic-ischemic encephalopathy)2-3 (neonatal convulsions in the fetus after childbirth),
2. Intracranial hemorrhage,
3. Apgar score < 4 at 5 minutes,
4. Arterial umbilical cord pH (potential of hydrogen) < 7.10,
5. Intrauterine fetal death, 6)intrapartal death.

Inclusion: All pregnancies in Stockholm with a fetus, born between 2014 and 2017 and without chromosomal abnormalities or other structural abnormalities, will be included in the project.

ELIGIBILITY:
Inclusion Criteria:

* All pregnancies in Stockholm with a fetus, born between 2014 and 2017 and without chromosomal abnormalities or other serious structural abnormalities, will be included in the project.

Exclusion Criteria:

* Pregnancies with known chromosomal abnormalities or other serious structural abnormalities

Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: All pregnant women in Stockholm during 2014-2017
Sampling Method: Probability Sample
Enrollment: 80000 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
The frequency of newborns with an affected perinatal outcome (low Apgar score and or affected acid-base status at labor) | 2014-2017
  Will the perinatal outcome at delivery( be measured as a low Apgar score at 5 minutes or an affected acid-base status in cord blood) be improved if IUGR(intrauterine growth restriction) is identified before labor

SECONDARY OUTCOMES:
The frequency of newborns with an affected perinatal outcome (low Apgar score and or affected acid-base status at labor)(2) | January 1th 2014- december 31th 2017
  Will the outcome changes persist if the group with IUGR will be divided into early- or late-diagnosed IUGR (before and after week 32 of pregnancy)?

CONTACTS AND LOCATIONS:
Overall Officials: Eva Wiberg-Itzel, PhD, Principal Investigator — Karolinska Institute Sodersjukhuset Sweden
Locations (1):
- Eva Wiberg-Itzel, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No